CLINICAL TRIAL: NCT06320509
Title: Interest of Urinary Oxygen Partial Pressure (PO2u) in Predicting the Onset or Recovery of Acute Renal Failure During Shock States - OXYpi Study
Acronym: OXYpi
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 49RC23_0417
Record Dates: First submitted 2024-02-27; First posted 2024-03-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Shock Circulatory
Keywords: Acute kidney injury; Continuous urine oxygen tension; Circulatory failure; Shock
MeSH Terms: conditions — Shock; Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shock population (Other): Insertion of bladder urine probe (Oxylite Pro ® device) and assessment of continuous uPO2
  Interventions: Biological: Continuous measurement of uPO2 (both groups)
- Without Shock Population (Other): Insertion of bladder urine probe (Oxylite Pro ® device) and assessment of continuous uPO2
  Interventions: Biological: Continuous measurement of uPO2 (both groups)

INTERVENTIONS:
Biological: Continuous measurement of uPO2 (both groups) — uPO2 is collected continuously for the first 5 days of admission or until discharge from intensive care or removal of the urinary catheter.

SUMMARY:
Shock state is defined as an acute, life-threatening, circulatory failure with impaired tissue oxygenation (or tissue hypoxia). The cause of the shock state can be septic, anaphylactic, hypovolemic or cardiogenic. Its management is based on etiological treatment and replacement of organ failures. Acute kidney injury (AKI) may be lead by renal hypoxia. Acute kidney injury is frequent in patients admitted to intensive care unit (ICU) and associated with an increased mortality. Serum creatinine is the reference biological marker in the diagnosis of Acute kidney injury. However, its use is limited by a delayed increase in plasma creatinine level in relation to the causal renal agression, at a time when renal tissue damage may already be established. Thus, the identification of a biological marker making it possible to estimate renal hypoxia continuously during a shock could allow us to identify early a situation at risk of evolving into Acute kidney injury.

The renal medulla is vulnerable to tissue hypoxia with a risk of acute tubular necrosis. As in situ measurement of mPO2 is not possible in current practice in humans, several studies have shown a positive correlation between variations in mPO2/uPO2 and occurence of Acute kidney injury. In humans, studies have shown a significant association between the reduction in uPO2 in cardiac surgeries and the occurrence of postoperative Acute kidney injury. The aim of the study is to describe the association between uPO2 values and the onset of Acute kidney injury and/or the ocurrence of early recovery of renal function after Acute kidney injury. Any patient in shock (group A) or without shock and requiring urinary catheterization as part of treatment (group B) admitted to the Medical-Intensive Care Unit of Angers University Hospital is eligible for inclusion. After inclusion, a continuous uPO2 measuring probe is introduced with the placement of the urinary probe. uPO2 is collected continuously for the first 5 days of admission or until discharge from intensive care or removal of the urinary catheter. uPO2 is also measured by a gasometry on a urine sample on a multi-daily basis. Serum creatinine is collected every 12 hours (twice a day) and diuresis every two hours for 5 days.

ELIGIBILITY:
Inclusion Criteria :

Group A:

- Patient admitted to Intensive Care Unit with a shock state defined by arterial hypotension requiring vascular filling and/or introduction of catecholamines - Age ≥ 18 years - Affiliated or benificiary of a social security scheme - Consent of the patient or a relative, or inclusion as part of an emergency inclusion procedure

Group B:

* Patient admitted to Intensive Care Unit without shock
* Requiring urinary catheterization as part of routine care
* Age ≥ 18 years
* Affiliated or benificiary of a social security scheme
* Consent of the patient or a relative, or inclusion as part of an emergency inclusion procedure

Exclusion Criteria:

- Preexisting chronic kidney disease (CKD) (GFR < 60 mL/min/1,73 m2 according to MDRD) - Chronic dialysis and/or kidney transplant - Anuria - Indication for renal replacement therapy (life-threatening hyperkaliemia, severe metabolic acidosis pH < 7,15, uremia > 40 mmol/L, pulmonary edema resistant to diuretics) - Patient requiring an extracorporeal life support (ECLS) - Pregnant, breastfeeding or parturient woman - Patient deprived of liberty by judicial or administrative decision - Patient under psychiatric care - Patient under legal protection measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2027-10-18 (Estimated); Study Completion 2028-01-18 (Estimated)

PRIMARY OUTCOMES:
A - For patients without acute kidney injury at inclusion, the occurence of acute kidney injury and its severity according to the KDIGO criteria | During the first 5 days after inclusion.
  A KDIGO Criteria: Increase in serum creatinine ≥ 26.5 µmol/L during the 48 hours following inclusion Or an increase of ≥ 1.5 fold the admission serum creatinine during the first 5 days Or Diuresis < 0.5 mL/kg/h for 6 hours during the first 5 days
B - For patients with acute kidney injury occurring during the first 3 days following inclusion, early recovery is defined by the return to pre-shock renal function 48 hours from the start of acute kidney injury | During the first 5 days after inclusion.
  A KDIGO Criteria: Increase in serum creatinine ≥ 26.5 µmol/L during the 48 hours following inclusion Or an increase of ≥ 1.5 fold the admission serum creatinine during the first 5 days Or Diuresis < 0.5 mL/kg/h for 6 hours during the first 5 days
C - For patients with acute kidney injury occurring at inclusion, describe the evolution of PO2u values in patients with worsening renal function | During the first 5 days after inclusion.
  A KDIGO Criteria: Increase in serum creatinine ≥ 26.5 µmol/L during the 48 hours following inclusion Or an increase of ≥ 1.5 fold the admission serum creatinine during the first 5 days Or Diuresis < 0.5 mL/kg/h for 6 hours during the first 5 days

SECONDARY OUTCOMES:
In patients in group A, assess the association between uPO2 variation and acute kidney injury, defined by KDIGO criteria, in different subgroups (septic shock, sepsis without norepinephrine, non-septic shock). | During the first 5 days after inclusion.
  KDIGO Criteria: Increase in serum creatinine ≥ 26.5 µmol/L during the 48 hours following inclusion Or an increase of ≥ 1.5 fold the admission serum creatinine during the first 5 days Or Diuresis < 0.5 mL/kg/h for 6 hours during the first 5 days.
  Sepsis is defined as a life-threatening organ dysfunction caused by suspected or confirmed infection.
  Septic shock is defined as a sepsis with need of norepinephrine.
In patients in group A with newly occured acute kidney injury, assess the association between uPO2 variation and recovery of acute kidney injury in different subgroups (septic shock, sepsis without norepinephrine, non-septic shock). | During the first 5 days after inclusion.
  For patients with acute kidney injury occurring during the first 3 days following inclusion, early recovery is defined by the return to pre-shock renal function 48 hours from the start of acute kidney injury.
  Sepsis is defined as a life-threatening organ dysfunction caused by suspected or confirmed infection.
  Septic shock is defined as a sepsis with need of norepinephrine.
In patients in group A, assess the evolution of uPO2 during the first 5 days in patients with and without sepsis | During the first 5 days after inclusion or until discharge from intensive care or removal of the urinary catheter.
  uPO2 is collected continuously for the first 5 days of admission or until discharge from intensive care or removal of the urinary catheter.
Describe the variation of uPO2 according to evolution of Mean Arterial Pressure and cardiac output in the subgroup of patients who received fluid expansion | During the first 5 days after inclusion or until discharge from intensive care or removal of the urinary catheter.
  uPO2 is collected continuously for the first 5 days of admission or until discharge from intensive care or removal of the urinary catheter.
  Mean Arterial Pressure is measured continuously with an in situ arterial line and cardiac output is measured invasively by transpulmonary thermodilution or a pulmonary arterial catheterization, or non-invasively by transthoraci echocardiography
Describe the variation of uPO2 according to evolution of Mean Arterial Pressure and cardiac output in the subgroup of patients who received blood transfusion | During the first 5 days after inclusion or until discharge from intensive care or removal of the urinary catheter.
  uPO2 is collected continuously for the first 5 days of admission or until discharge from intensive care or removal of the urinary catheter.
  Mean Arterial Pressure is measured continuously with an in situ arterial line and cardiac output is measured invasively by transpulmonary thermodilution or a pulmonary arterial catheterization, or non-invasively by transthoracic echocardiography
In patients with need of increasing Mean Arterial Pressure by increase of norepinephrine doses, describe the evolution of uPO2 according to Mean Arterial Pressure evolution. | During 1 hour from the beginning of the increase of norepinephrine doses.
  uPO2 is collected continuously for the first 5 days of admission or until discharge from intensive care or removal of the urinary catheter.
  Mean Arterial Pressure is measured continuously with an in situ arterial line.
In patients with need of introduction or increase of dobutamine, describe the evolution of uPO2 according to cardiac output or Mean Arterial Pressure evolution. | During 1 hour from the introduction or increase of dobutamine.
  uPO2 is collected continuously for the first 5 days of admission or until discharge from intensive care or removal of the urinary catheter.
  Mean Arterial Pressure is measured continuously with an in situ arterial line and cardiac output is measured invasively by transpulmonary thermodilution or a pulmonary arterial catheterization, or non-invasively by transthoraci echocardiography
Evaluation the correlation between uPO2 assessed by Oxylite Pro® device and urinary gasometry. | During the first 5 days after inclusion or until discharge from intensive care or removal of the urinary catheter.
  Evaluation the correlation between uPO2 assessed by Oxylite Pro® device and urinary gasometry.
In patients without shock, describe the evolution of uPO2 during the first 5 days. | During the first 5 days after inclusion or until discharge from intensive care or removal of the urinary catheter.
  uPO2 is collected continuously for the first 5 days of admission or until discharge from intensive care or removal of the urinary catheter.
In patients with septic shock, build up a biocollection, enabling further analyses to be carried out at a later date | During the first 5 days after inclusion or until discharge from intensive care or removal of the urinary catheter.
  Build up a biocollection by taking additional blood and urine samples
In patients who, during their treatment, have an indication for the introduction or increase of vasopressin: assess the impact of introducing/increasing vasopressin on PO2u. | During 20 minutes from the beginning of the increase of vasopressine doses
For patients whose skin recoloration time and PO2u are assessed before and after a procedure, describe the correlation between changes in PO2u and skin recoloration time during each procedure | During 1 hour from the beginning of the increase of norepinephrine doses, during 1 hour from the introduction or increase of dobutamine, during 20 minutes from the beginning of the increase of vasopressine doses

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - University Hospital of Angers, Angers
  - Bicêtre Hospital, Le Kremlin-Bicêtre

IPD SHARING:
Plan to Share IPD: No